CLINICAL TRIAL: NCT00556153
Title: [F-18]Fluoro-DOPA PET Imaging of Brain Tumors in Children
Status: Withdrawn | Type: Observational
Why Stopped: No participants ever enrolled.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CCHMC IRB# 04-09011
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Brain Tumors
Keywords: brain tumors, children
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Phase I: Children, ages 5-15 years with brain tumors
  Interventions: Drug: [F-18]Fluoro-DOPA PET, a diagnostic radiopharmaceutical

INTERVENTIONS:
Drug: [F-18]Fluoro-DOPA PET, a diagnostic radiopharmaceutical — A single dosage of the diagnostic drug will be administered to individuals who meet inclusion criteria after informed consent.

SUMMARY:
The first phase of the study will investigate if there is increased uptake of [F-18]FDOPA in pediatric brain tumors when compared to normal brain tissue.

DETAILED DESCRIPTION:
The first phase of the study will investigate if there is increased uptake of [F-18]FDOPA in pediatric brain tumors when compared to normal brain tissue. Tne subjects between ages 5 and 17 years will be studies, to determine if there is increased uptake of [F-18]FDOPA in pediatric brain tumors when compared to normal brain tissue. Drug safety will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Documented brain tumor at diagnosis or relapse, including high grade glioma, low grade glioma, medulloblastoma including PNET, optic pathway glioma, brainstem glioma, ependymoma.

Exclusion Criteria:

* Pregnancy
* Requirement for sedation
* Lack of informed consent

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 5-15 years, with brain tumors
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Increased uptake of [F-18]FDOPA in pediatric brain tumors compared to contralateral normal brain tissue as measured by standardized uptake value and tumor/non-tumor uptake ratios | 15-30 minutes after IV administration

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Gelfand, M.D., Principal Investigator — Cincinnati Children's Hospital, Cincinnati, OH